CLINICAL TRIAL: NCT05686590
Title: Prehospital Provider Training Using Augmented Reality Simulation: A Mixed-Methods Study
Brief Title: Prehospital Provider Training With Augmented Reality (AR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Caruso (Other)
Responsible Party: Sponsor-Investigator, Thomas Caruso, Clinical Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 67544
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Hypoglycemia; Pediatric ALL
MeSH Terms: conditions — Hypoglycemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Augmented Reality Enhanced Simulation (Treatment group) (Experimental): Each simulation will have between two and five participants. After consent, demographic data will be collected. Then, a study RA will fit a Magic Leap One (ML1) headsets (Magic Leap Inc., Plantation, FL) to participants. Following a scripted briefing, the instructor will also orient the participants to the ML1 headset for those in that group. After orienting the participant to the use of the headsets, the instructor will remain in a room separate from the participants, who will conduct the scenario outside. This will enable assessment of the feasibility of providing simulation instruction remotely. Prior to starting the scenario, the simulation instructor will conduct an orientation to review the core tenets of effective communication skills during prehospital care.
  Interventions: Behavioral: Augmented Reality Headset

INTERVENTIONS:
Behavioral: Augmented Reality Headset — The simulation scenario will be a pediatric hypoglycemia-induced seizure case, which will be done through an AR simulation. AR (Augmented Reality) headset, which is a device that the participants will wear over their head and eyes and will add holographic elements to a live view of workplace training scenario.

SUMMARY:
The goal is to evaluate the acceptance of Augmented Reality (AR) simulation as a learning modality for prehospital providers. The simulation itself is grounded in traditional best practices for simulation delivery and design as well as prior literature on simulation training for prehospital providers; the focus of this study is the participants' experiential interaction with AR and the simulation resources.

ELIGIBILITY:
Inclusion Criteria:

* Trainees/ faculty working and/or volunteering at LPCH/SHC facilities as well as community based prehospital providers
* 18 years and older

Exclusion Criteria:

* Participants who do not consent
* Have a history of severe motion sickness
* Currently have nausea
* History of seizures
* Are clinically unstable
* Currently using corrective glasses (not compatible with AR headset)
* Currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Thematic Analysis of Post-Simulation Discussions | Duration of post-simulation debrief (15-20 minutes)
  The primary aim is to study the acceptance of AR simulation amongst prehospital providers via thematic analysis of semi-structured discussions using qualitative research methods.

SECONDARY OUTCOMES:
System Usability Scale (SUS) | Duration of Intervention (less than one hour)
  The first secondary aim is to evaluate AR simulation usability amongst prehospital providers via the System Usability Scale (SUS).
Headset Ergonomics | Duration of Intervention (less than one hour)
  The final secondary aim will evaluate the ergonomics of the headset via the ISO 9241-400 assessment of human-ergonomic factors.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Mountain View Fire Department, Mountain View, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California

IPD SHARING:
Plan to Share IPD: No